CLINICAL TRIAL: NCT06741683
Title: A Randomized, Double-Blind, Placebo-Controlled (Participants Aged 18 to 60 Years) and Open-Label (Participants Aged 4 to 17 Years), Phase 2/3 Trial to Evaluate the Immunogenicity and Safety of 2 Doses of a Dengue Tetravalent Vaccine (Live, Attenuated) (TDV) Administered Subcutaneously to Healthy Adults, Adolescents, and Children in Japan
Brief Title: A Study of Dengue Tetravalent Vaccine (TDV) in Healthy Participants in Japan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DEN-324; 2024-000341-27 (EudraCT Number); jRCT2071240088 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Cohort 1 is randomized and double-blinded. Cohort 2 is non-randomized and open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: TDV 0.5 mL (Experimental): Participants with the age group 18 to 60 years will receive TDV, 0.5 milliliter (mL) subcutaneous (SC) injections, on Day 1 and Day 90.
  Interventions: Biological: TDV
- Cohort 1: Placebo (Placebo Comparator): Participants with the age group 18 to 60 years will receive placebo (normal saline), 0.5 mL SC injections, on Day 1 and Day 90.
  Interventions: Other: Placebo
- Cohort 2: TDV 0.5 mL (Experimental): Participants with the age group 4 to 17 years will receive TDV, 0.5 mL SC injections, on Day 1 and Day 90.
  Interventions: Biological: TDV

INTERVENTIONS:
Biological: TDV — TDV SC injection.
  Other Names: TAK-003
  Arms: Cohort 1: TDV 0.5 mL; Cohort 2: TDV 0.5 mL
Other: Placebo — Placebo SC injection.
  Other Names: Placebo SC injection.
  Arms: Cohort 1: Placebo

SUMMARY:
Dengue fever is caused by an infection with the dengue virus. Vaccination with TDV can help prevent dengue fever.

The main purpose of this study is to learn about TDV's ability to create an immune response in adults, adolescents, and children administered. In this study, participants will receive 2 vaccinations with TDV (the second 3 months after the first). During the study, participants will visit their study clinic 5 times.

Participants will be in this study for approximately 270 days (9 months).

ELIGIBILITY:
Inclusion Criteria:

1. Participant aged >=4 to less than or equal to (<=) 60 years at the time of signing the informed consent/pediatric assent form.
2. Participant is Japanese male or female.
3. Participant is in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator.
4. Participant and/or the participant's legally acceptable representative (LAR) who have signed and dated a written, informed consent/pediatric assent form, and any required privacy authorization prior to the initiation of any trial procedures, and after the nature of the trial has been explained.
5. Participant can comply with trial procedures and is available for the duration of follow-up.

Exclusion Criteria:

1. Participant has contraindication(s), warning(s), and/or precaution(s) applicable to vaccination with TDV as specified in the Investigator's Brochure.
2. Participant has a known hypersensitivity or allergy to any of the IMP components (including excipients of the IMP).
3. Participant has behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the trial.
4. Participant has a history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (example, Guillain-Barré syndrome).
5. Participant has a clinically significant active infection (as assessed by the investigator) or body temperature greater than (>) 38.0 degrees Celsius (°C) (>100.4 degrees Fahrenheit [°F]) within 3 days of intended IMP administration on Day 1 (Month [M] 0).

   Note: In principle, oral temperature should be measured for body temperature. In cases where it is difficult to measure oral temperature, such as in young children, underarm (axillary) temperature may be used instead.
6. Participant has an illness, or history of any illness that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the participant due to involvement in this trial.
7. Participant has a known or suspected impairment/alteration of immune function, including:

   1. Chronic administration of oral and/or parenteral steroids at doses considered sufficiently immunosuppressive (example, >=2 milligram per kilogram [mg/kg] body weight prednisone [or equivalent] for >=14 consecutive days, or >=20 milligram per day [mg/day] prednisone [or equivalent] administered for >=14 consecutive days) within 60 days prior to Day 1 (M0), Note: use of corticosteroids by inhaled, intranasal, intra-articular, bursal, tendon injection, or topical routes is allowed.
   2. Receipt of blood, immunoglobulins, blood products, and/or plasma derivatives within the 90 days prior to Day 1 (M0).
   3. Receipt of immunostimulants within 60 days prior to Day 1 (M0).
   4. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (M0).
   5. Reported or known symptomatic HIV infection or asymptomatic HIV infection when accompanied by evidence of impaired immune function.
   6. Reported or known Hepatitis B and/or Hepatitis C virus infection.
   7. Genetic immunodeficiency.
8. Participant has known or suspected abnormalities of splenic or thymic function.
9. Participant has a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
10. Participant has a serious chronic or progressive disease deemed to be preclusive to trial entry, that is not medically stable according to the judgment of the investigator.
11. Participant is participating in any clinical trial with another investigational product within 30 days prior to Day 1 (M0) or plans to participate in another clinical trial at any time during the conduct of this trial.
12. Participant has previously received a vaccination against flavivirus other than Japanese encephalitis (JE) (investigational or licensed).
13. Participant who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to Day 1 (M0) or who are planning to receive any vaccine other than IMP within 28 days of IMP administration.
14. Participant who received a coronavirus vaccine within 14 days prior to Day 1 (M0).
15. Participant who received a vaccine authorized for emergency use within 28 days prior to Day 1 (M0).
16. Participant who received any JE vaccines within 28 days prior to Day 1 (M0) or who are planning to receive any JE vaccines during the trial period.
17. Previous participation in any clinical trial of a dengue or other flavivirus candidate vaccine, except for participants who received placebo in those trials.
18. Participant with body mass index (BMI) >=35 kilograms per square meter (kg/m^2) on Day 1 (M0).
19. Participant who intends to travel to dengue endemic areas during the trial period.
20. Participant with documented or suspected disease caused by a flavivirus and participants with a history of prolonged (>=1 year) habitation in a dengue endemic area.
21. Participant with history of substance or alcohol abuse within the past 2 years prior to Day 1 (M0).
22. Female participants who are pregnant (that is, a positive or indeterminate pregnancy test) or breastfeeding.
23. Females of childbearing potential who are sexually active and who have not used any of the acceptable contraceptive methods for at least 2 months prior to Day 1 (M0).

    1. "Childbearing potential" is defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy.
    2. Acceptable contraceptive methods" are defined as one or more of the following:

       * Hormonal contraceptive.
       * Barrier method (condom or diaphragm) every time during intercourse.
       * Intrauterine device.
       * Monogamous relationship with a vasectomized partner. The partner must have been vasectomized for at least 6 months prior to the participant's trial enrollment.
24. Females of "childbearing potential" or non-sterilized males, who refuse to use an "acceptable contraceptive method" up to 6 weeks post second IMP administration on Day 90 (M3). In addition, they must be advised not to donate ova or sperm during this period.
25. A first degree relative is involved in the conduct of this trial.

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 187 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Percentage of Seropositive Participants for Each of the 4 Dengue Virus Serotypes on Day 120 | Day 120
  Seropositivity is defined as a reciprocal neutralizing titer greater than or equal to (>=) 10. The 4 dengue virus serotypes (DENV) are DENV-1, DENV-2, DENV-3 and DENV-4.

SECONDARY OUTCOMES:
Percentage of Seropositive Participants for Each of the 4 Dengue Virus Serotypes on Day 1, Day 30, Day 90 and Day 270 | Day 1, Day 30, Day 90 and Day 270
  Seropositivity is defined as a reciprocal neutralizing titer >=10. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Virus Serotypes on Day 1, Day 30, Day 90, Day 120 and Day 270 | Day 1, Day 30, Day 90, Day 120 and Day 270
  GMTs of neutralizing antibodies will be measured by microneutralization Test (MNT) for each of the 4 Dengue serotypes. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Percentage of Seropositive Participants for Multiple (2, 3, or 4) Dengue Serotypes on Day 1, Day 30, Day 90, Day 120 and Day 270 | Day 1, Day 30, Day 90, Day 120 and Day 270
  Seropositivity is defined as a reciprocal neutralizing titer >=10 for multiple dengue serotypes (2, 3, or 4).
Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 days After Vaccination at Day 1 and Day 90 | For 7 days after vaccination at Day 1 and Day 90
  The solicited local (at injection site) AEs includes pain, erythema, and swelling.
Number of Participants with Solicited Local (Injection Site) AEs by Severity for 7 days After Vaccination at Day 1 and Day 90 | For 7 days after vaccination at Day 1 and Day 90
  The solicited local (at injection site) AEs includes pain, erythema, and swelling. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Number of Participants With Solicited Systemic AEs for 14 days After Vaccination at Day 1 and Day 90 | For 14 days after vaccination at Day 1 and Day 90
  The solicited systemic AEs for less than (<) 6 years of age will be fever, irritability/fussiness, drowsiness, and loss of appetite; and for >=6 years of age will be asthenia, fever, headache, malaise, and myalgia.
Number of Participants With Solicited Systemic AEs by Severity for 14 days After Vaccination at Day 1 and Day 90 | For 14 days after vaccination at Day 1 and Day 90
  The solicited systemic AEs for <6 years of age will be fever, irritability/fussiness, drowsiness, and loss of appetite; and for >=6 years of age will be asthenia, fever, headache, malaise, and myalgia. The AEs will be graded by investigator as Grade 0: none, Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants With Any Unsolicited AEs for 28 days After Vaccination at Day 1 and Day 90 | For 28 days after vaccination at Day 1 and Day 90
  An unsolicited AE is any AE reported by the participant that is not specified as a solicited AE or is specified as a solicited AE but starts outside the period for reporting a solicited AE (that is, 7 days and 14 days in total including the day of Investigational Medicinal Product [IMP] administration).
Percentage of Participants With Serious Adverse Event (SAE) | From first vaccination on Day 1 through the end of trial (up to Day 270)
  A SAE is defined as any untoward medical occurrence that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/ incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, is an important medical event.
Percentage of Participants With Medically Attended AEs (MAAEs) | From first vaccination on Day 1 through the end of trial (up to Day 270)
  MAAEs are defined as AEs leading to an unscheduled visit or by a healthcare professional including visits to an emergency department (medically attended visits), but not fulfilling seriousness criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- Japan (5):
  - PS Clinic, Fukuoka, Fukuoka
  - Saitama City Hospital, Saitama-shi, Saitama
  - Sumida Hospital, Sumida-ku, Tokyo
  - OKURA Otolaryngology Clinic, Toshima-ku, Tokyo
  - Tamura Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/f23b144ad81e40b4